CLINICAL TRIAL: NCT04348448
Title: Observational Study on the Use of Canakinumab Administered Subcutaneously in the Treatment of Patients With COVID-19 Pneumonia
Brief Title: Observational Study, Use of Canakinumab Administered Subcutaneously in the Treatment COVID-19 Pneumonia
Status: Terminated | Type: Observational
Why Stopped: due to covid
Sponsor: AUSL Romagna Rimini (Other)
Responsible Party: Sponsor
Other Study IDs: CANASCOV
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — canakinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Canakinumab 150 MG/ML [Ilaris] — COVID-19

SUMMARY:
The study is configured as a retrospective and prospective observational study. The study will be multi-center and will involve all COVID-19 pneumonia patients treated with canakinumab administered subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

* patients with COVID 19 who have received or are candidates to receive treatment with canakinumab subcutaneously
* Age> 18 years
* Pneumonia diagnosed with Chest X-ray / or Chest CT

Exclusion Criteria:

* Patients with Covid19-related pathology in the context of another cause of major admission (trauma, surgery)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with COVID 19
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
intensive care treatment | 9 months
  percentage of patients treated with canakinumab sc who do not require intensive care treatment during hospitalization for COVID-19

SECONDARY OUTCOMES:
ICU stay times | 9 months
  ICU stay times
% died after 1 month after treatment | 9 months
  percentage of patients who died 1 month after treatment
hospitalization | 9 months
  time of hospitalization
adverse event | 9 months
  number of adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Ausl della Romagna, Ravenna, Italy